CLINICAL TRIAL: NCT05716529
Title: Functional Outcomes of a Criterion-based Rehabilitation Protocol for Anterior Cruciate Ligament Reconstruction in Amateur Athletes: a Randomized Clinical Trial
Brief Title: Functional Outcomes of an Accelerated Rehabilitation Protocol for ACL Reconstruction in Amateur Athletes
Acronym: ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Lecturer of Orthopedics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 004257
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: ACL Injury; Rehabilitation After ACL Reconstruction; Accelerated Protocol
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accelerated rehabilitation protocol (Experimental): It's a four phases rehabilitation protocol mainly based on the remodeling process of the graft., emphasizing full passive knee extension, immediate weight bearing as tolerated and functional exercises
  Interventions: Other: rehabilitation protocol
- conventional physical therapy program (Active Comparator): Current conventional protocols were based mainly on biological tissue healing time frames. These protocols emphasize pain reduction, full passive knee extension, quadriceps strength training, immediate motion, immediate par¬tial weight bearing (only if there is a correct gait pattern without any complications), and functional exercises
  Interventions: Other: rehabilitation protocol

INTERVENTIONS:
Other: rehabilitation protocol — It's a four phases rehabilitation protocol mainly based on the remodeling process of the graft., emphasizing full passive knee extension, immediate weight bearing as tolerated and functional exercises

SUMMARY:
The main goal of a rehabilitation program after an ACL reconstruction is to regain mobility and muscle function and ultimately to return to sports participation. Purpose of the study: to investigate the effect of the accelerated rehabilitation program on knee pain, and function in patients post ACLR surgery. Fifty adult amateur males athletes who underwent ACLR surgery participated in this study, their age ranged from 18 to 35years.They were randomly assigned into two equal groups. Group (A) received accelerated rehabilitation protocol and group (B) received conventional physical therapy program. Treatment sessions were conducted 5 times per week for 22 weeks for both groups. All patients assessed pre and post treatment for pain intensity using visual analogue scale (VAS), and knee function using knee injury and osteoarthritis outcome score (KOOS), knee effusion, and LSI of Hop test.

ELIGIBILITY:
Inclusion Criteria:

* Patients were participated in this study if they fulfilled the following criteria:

  * Underwent pre-operative rehabilitation program with minimal knee effusion and full extension, good patellofemoral mobility, and the patient can actively control the quadriceps.
  * Have an ACLR with an autolongous hamstring (HT) graft.
  * Age range from 18-40 years old.
  * Football players or who perform physically demanding work.
  * Have no other ligamentous injury.
  * Have nomeniscectomy previous to or simultaneouswith ACLR.
  * Have no cartilage damage.

Exclusion Criteria:

* • Patients younger than 18 or older than 35 years old

  * Have ACLR with any graft other than hamstring (HT) graft
  * Have ACL revision surgery
  * Have other ligamentous injury
  * Have a meniscectomy previous to or simultaneous with ACLR.
  * Had meniscal repair simultaneously with ACLR
  * Have cartilage damage.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 22 weeks
  It is a 100-mm horizontal line anchored by word descriptors at each end by ""no pain"" on the left and ""worst imaginable pain"" on the right

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 22 weeks
  it is a 42-item self-questionnaire with five subscales. A five-point scale ranging from 0 (no problem) to 4 (extreme problems) was used to score each item and the scores of each subscale were individually transformed into a 0-100 scale (0 = extreme knee problems, 100 = no knee problem)
limb symmetry index of Hop test battery | 22 weeks
  The mean score of the results of each item of hop test battery of the injured limb was divided by the corresponding mean score of the uninjured limb and the result was multiplied by 100. Hop test battery consists of the following: (1) vertical jump, (2) hop for distance, (3) drop jump followed by a double hop for distance, (4) square hop and (5) side hop
knee effusion grading scale | 22 weeks
  It"s a reliable and valid method which Based on a stroke test, where effusion of the knee joint is quantified using a 5-point scale. A 0 grade means no wave is produced with the downward stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university, Gamasa, Eldakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No